CLINICAL TRIAL: NCT05747937
Title: Longitudinal Assessment of Autonomic and Sensory Nervous System in ALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SBLAB/SLA20
Record Dates: First submitted 2023-01-26; First posted 2023-02-28 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Autonomic nervous system; skin biopsy; biomarkers; cutaneous sensory an autonomic innervation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Masking Description: There are not masking participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amyotrophic Lateral Sclerosis patients (Experimental): Amyotrophic Lateral Sclerosis (ALS) patients within 18 months from symptoms onset will be recruited
  Interventions: Diagnostic Test: Skin biopsy; Diagnostic Test: Cardiovascular Reflexes testing; Diagnostic Test: Administration of clinical scales evaluating autonomic symptoms, pain small fiber neuropathy symptoms; Diagnostic Test: Dinamic Sweat Test
- Healthy controls (Active Comparator): A population of healthy controls matched for sex and age will be enrolled
  Interventions: Diagnostic Test: Skin biopsy; Diagnostic Test: Cardiovascular Reflexes testing; Diagnostic Test: Administration of clinical scales evaluating autonomic symptoms, pain small fiber neuropathy symptoms; Diagnostic Test: Dinamic Sweat Test

INTERVENTIONS:
Diagnostic Test: Skin biopsy — A punch skin biopsy of 3mm will be used to analyze cutaneous innervation
Diagnostic Test: Cardiovascular Reflexes testing — Cardiovascular reflex tests including deep breathing, head-up Tilt, standing, isometric exercises, mental arithmetic and Valsalva maneuver.
Diagnostic Test: Administration of clinical scales evaluating autonomic symptoms, pain small fiber neuropathy symptoms — We'll characterize patients' symptoms through the administration of clinical scales such as: SCOPA-AUT autonomic symptoms scale; Brief Pain Inventory questionnaire
Diagnostic Test: Dinamic Sweat Test — Test for the functional assessment of postganglionic sudomotor pathway

SUMMARY:
The goal of this interventional non-pharmacological study is to evaluate, using a multimodal approach, the progression of autonomic and sensory involvement in in amyotrophic lateral sclerosis (ALS) patients enrolled within 18 months from motor onset and its relationship with the progression of overall clinical disability.

The main questions it aims to answer are:

* Is autonomic dysfunction at diagnosis associated with disease progression and survival in patients with Amyotrophic Lateral Sclerosis ?
* Can we identify in the skin biomarkers to be used as reliable measures of disease progression and to apply in future clinical trials for patient stratification and to assess response to drug treatment ? Participants at time 0 will receive a full clinical and instrumental examination and a blood sample testing to check inclusion and exclusion criteria, genetic screening for the most common genes associated with ALS (SOD1, FUS, TARDBP and c9orf72), questionnaires about clinical characteristics, quality of life, pain and a multidomain battery of neuropsychological tests, multimodal assessment of the autonomic nervous system including skin biopsy for morphological study. At follow-up we'll perform clinical scales and skin biopsy.

Researchers will compare results from ALS patients with data obtained from a population of age and sex matched healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* ALS patients will be recruited within 18 months from the motor symptoms onset

Exclusion Criteria:

* glucose intolerance or conditions potentially affecting the peripheral nervous system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensory peripheral innervation (IENF) | At recruitment
  Quantification Intraepidermal Nerve Fibers (IENF ff/mm) in skin biopsy from fingertip, thigh and leg.
Autonomic peripheral innervation | At recruitment
  Quantification of nerves in sweat gland (fiber lenght/um3) in skin biopsy from fingertip, thigh and leg.
  Quantification of nerves in arrector pili muscle (ff/mm) in skin biopsy from thigh and leg.
Autonomic peripheral innervation | At follow-up, an average of 6 months
  Quantification sweat gland (fiber lenght/um3) and arrector pili muscle (ff/mm) innervation in skin biopsy from thigh.
Sensory peripheral innervation (IENF) | At follow-up, an average of 6 months
  Quantification Intraepidermal Nerve Fibers (IENF ff/mm) in skin biopsy from thigh.

SECONDARY OUTCOMES:
Sensory and autonomic symptoms evaluated by clinical scales | At the recruitment
  Data of sensory and autonomic symptoms (Small fiber neuropathy Symptoms inventory questionnaire (SFN-SIQ) and Scale for Outcomes in Parkinson's disease for Autonomic Symptoms (SCOPA AUT)) will be collected
Sensory and autonomic symptoms evaluated by clinical scales | At follow-up, an average of 6 months
  Data of sensory and autonomic symptoms (Small fiber neuropathy Symptoms inventory questionnaire (SFN-SIQ) and Scale for Outcomes in Parkinson's disease for Autonomic Symptoms (SCOPA AUT)) will be collected
Assessment of Cardiovascular function | baseline
  Data from cardiovascular reflex test will be analyzed and compared with morphological data and clinical motor severity
Sudomotor function | baseline
  Data from dinamic sweat test will be analyzed and compared with morphological data and clinical motor severity

CONTACTS AND LOCATIONS:
Overall Officials: Maria Nolano, MD, PhD, Principal Investigator — Istituti Clinici Scientifici Maugeri SpA
Locations (2):
- Italy (2):
  - ICS Maugeri - IRCCS of Telese Terme, Telese Terme, Benevento
  - Department of Neurosciences, Reproductive Sciences and Odontostomatology, University of Naples Federico II, Napoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahoney CJ, Ahmed RM, Huynh W, Tu S, Rohrer JD, Bedlack RS, Hardiman O, Kiernan MC. Pathophysiology and Treatment of Non-motor Dysfunction in Amyotrophic Lateral Sclerosis. CNS Drugs. 2021 May;35(5):483-505. doi: 10.1007/s40263-021-00820-1. Epub 2021 May 15. PMID 33993457
- [Background] Gentile F, Scarlino S, Falzone YM, Lunetta C, Tremolizzo L, Quattrini A, Riva N. The Peripheral Nervous System in Amyotrophic Lateral Sclerosis: Opportunities for Translational Research. Front Neurosci. 2019 Jun 25;13:601. doi: 10.3389/fnins.2019.00601. eCollection 2019. PMID 31293369
- [Background] Sassone J, Taiana M, Lombardi R, Porretta-Serapiglia C, Freschi M, Bonanno S, Marcuzzo S, Caravello F, Bendotti C, Lauria G. ALS mouse model SOD1G93A displays early pathology of sensory small fibers associated to accumulation of a neurotoxic splice variant of peripherin. Hum Mol Genet. 2016 Apr 15;25(8):1588-99. doi: 10.1093/hmg/ddw035. Epub 2016 Feb 9. PMID 26908600
- [Background] Weis J, Katona I, Muller-Newen G, Sommer C, Necula G, Hendrich C, Ludolph AC, Sperfeld AD. Small-fiber neuropathy in patients with ALS. Neurology. 2011 Jun 7;76(23):2024-9. doi: 10.1212/WNL.0b013e31821e553a. PMID 21646630
- [Background] Truini A, Biasiotta A, Onesti E, Di Stefano G, Ceccanti M, La Cesa S, Pepe A, Giordano C, Cruccu G, Inghilleri M. Small-fibre neuropathy related to bulbar and spinal-onset in patients with ALS. J Neurol. 2015;262(4):1014-8. doi: 10.1007/s00415-015-7672-0. Epub 2015 Feb 17. PMID 25683764
- [Background] Nolano M, Provitera V, Manganelli F, Iodice R, Caporaso G, Stancanelli A, Marinou K, Lanzillo B, Santoro L, Mora G. Non-motor involvement in amyotrophic lateral sclerosis: new insight from nerve and vessel analysis in skin biopsy. Neuropathol Appl Neurobiol. 2017 Feb;43(2):119-132. doi: 10.1111/nan.12332. Epub 2016 Jul 7. PMID 27288647
- [Background] deCarvalho M, Gromicho M, Andersen P, Grosskreutz J, Kuzma-Kozakiewicz M, Petri S, Uysal H, Pinto S. Peripheral neuropathy in ALS: phenotype association. J Neurol Neurosurg Psychiatry. 2021 Oct;92(10):1133-1134. doi: 10.1136/jnnp-2020-325164. Epub 2020 Dec 28. No abstract available. PMID 33372053
- [Background] Chio A, Mora G, Lauria G. Pain in amyotrophic lateral sclerosis. Lancet Neurol. 2017 Feb;16(2):144-157. doi: 10.1016/S1474-4422(16)30358-1. Epub 2016 Dec 8. PMID 27964824
- [Background] Fasolino A, Di Stefano G, Leone C, Galosi E, Gioia C, Lucchino B, Terracciano A, Di Franco M, Cruccu G, Truini A. Small-fibre pathology has no impact on somatosensory system function in patients with fibromyalgia. Pain. 2020 Oct;161(10):2385-2393. doi: 10.1097/j.pain.0000000000001920. PMID 32897040
- [Background] Finnerup NB, Haroutounian S, Kamerman P, Baron R, Bennett DLH, Bouhassira D, Cruccu G, Freeman R, Hansson P, Nurmikko T, Raja SN, Rice ASC, Serra J, Smith BH, Treede RD, Jensen TS. Neuropathic pain: an updated grading system for research and clinical practice. Pain. 2016 Aug;157(8):1599-1606. doi: 10.1097/j.pain.0000000000000492. PMID 27115670
- [Background] Damon-Perriere N, Foubert-Samier A, De Cock VC, Gerdelat-Mas A, Debs R, Pavy-Le Traon A, Senard JM, Rascol O, Tison F, Meissner WG. Assessment of the Scopa-Aut questionnaire in multiple system atrophy: relation to UMSARS scores and progression over time. Parkinsonism Relat Disord. 2012 Jun;18(5):612-5. doi: 10.1016/j.parkreldis.2011.12.009. Epub 2012 Jan 9. PMID 22236582
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847